CLINICAL TRIAL: NCT02678351
Title: 68Ga-PSMA-11 PET/MRI for Detection of Regional Nodal and Distant Metastases in Patients With Intermediate and High-Risk Prostate Cancer
Brief Title: 68Ga-PSMA-11 PET/MRI in Finding Tumors in Patients With Intermediate or High-Risk Prostate Cancer Undergoing Surgery
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Andrei Iagaru (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Andrei Iagaru, Associate Professor of Radiology, Stanford University
Organization: Stanford University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB-35931; NCI-2016-00092 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); PROS0075 (Other: OnCore ID)
Record Dates: First submitted 2016-02-02; First posted 2016-02-09 (Estimated); Results first posted 2022-03-04 (Actual); Last update posted 2022-03-04 (Actual); Status verified 2022-03

CONDITIONS: Stage II Prostate Adenocarcinoma; Stage III Prostate Adenocarcinoma
MeSH Terms: interventions — gallium 68 PSMA-11; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 68Ga-PSMA PET/MRI (Experimental): Patients receive 68Ga-PSMA-11 IV. Patients then undergo PET/MRI after 45 minutes of administration of radiopharmaceutical injection.
  Interventions: Drug: 68Ga-PSMA-11; Procedure: Magnetic resonance imaging (MRI); Procedure: Positron Emission Tomography (PET)

INTERVENTIONS:
Drug: 68Ga-PSMA-11 — Undergo 68Ga-PSMA-11 PET/MRI
  Other Names: 68-gallium prostate-specific membrane antigen 11 positron emission tomography/magnetic resonance imaging; HBED CC PSMA; DFKZ 11; Heidelberg compound
Procedure: Magnetic resonance imaging (MRI) — Undergo 68Ga-PSMA-11 PET/MRI
  Other Names: Nuclear magnetic resonance imaging; MRI imaging; NMR Imaging; NMRI
Procedure: Positron Emission Tomography (PET) — Undergo 68Ga-PSMA-11 PET/MRI
  Other Names: PET scan; Positron Emission Tomography Scan; Proton magnetic resonance spectroscopic imaging

SUMMARY:
This phase 2-3 trial studies the utility of 68-gallium (68Ga)-prostate-specific membrane antigen 11 (PSMA-11) positron emission tomography/magnetic resonance imaging (PET/MRI) to find tumors in patients with prostate cancer who are undergoing resection surgery for prostate cancer that is prognostically expected to spread quickly (intermediate-risk) or is likely to come back or spread (high-risk). Diagnostic procedures, such as PET/MRI, may help find and diagnose prostate cancer, and reveal out how far the disease has spread. Radioactive drugs, such as 68Ga-PSMA-11, may bind to tumor cells that have specific receptors, and may allow doctors to see smaller tumors than the standard of care contrast-enhanced computed tomography (CT) or MRI scan.

DETAILED DESCRIPTION:
OBJECTIVES:

1. To evaluate 68Ga-PSMA-11 PET/MRI for detection of tumor metastases in patients with intermediate and high-risk prostate cancer scheduled to undergo prostatectomy with lymph node dissection.
2. To assess sensitivity (positive predictive value) and specificity (negative predictive value) of 68Ga-PSMA-11 PET/MRI for the detection of regional nodal metastases compared to pathology at radical prostatectomy.

OUTLINE:

Participants will receive 68Ga-PSMA-11 intravenously (IV). Patients then undergo PET/MRI after 45 minutes of administration of radiopharmaceutical injection.

After completion of study, patients are followed up at 24 to 48 hours.

ELIGIBILITY:
INCLUSION CRITERIA

* Biopsy-proven prostate adenocarcinoma
* Planned prostatectomy with lymph node dissection
* Intermediate- to high-risk disease (as determined by elevated prostate-specific antigen (PSA) [PSA > 10], T stage [T2b or greater], Gleason score [Gleason score > 6] or other risk factors)
* Karnofsky performance status of ≥ 50 [or Eastern Cooperative Oncology Group (ECOG)/World Health Organization (WHO) equivalent]
* Diagnostic CT or MRI performed within 90 days of the research PET
* Able to provide written consent

ExCLUSION CRITERIA

* Patients not capable of getting PET study due to weight, claustrophobia, or inability to lay still for the duration of the exam
* Neoadjuvant chemotherapy or radiation therapy prior to prostatectomy, including focal ablation techniques (HiFu)
* Androgen deprivation therapy or other neoadjuvant treatments prior to PET imaging and surgery
* Metallic implants (contraindicated for MRI)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2016-04-18 (Actual); Primary Completion 2020-12-13 (Actual); Study Completion 2021-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrei Iagaru, Principal Investigator — Stanford University
Locations (1):
- Stanford University, School of Medicine, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Duan H, Baratto L, Hatami N, Liang T, Levin CS, Khalighi MM, Iagaru A. Reduced Acquisition Time per Bed Position for PET/MRI Using 68Ga-RM2 or 68Ga-PSMA-11 in Patients With Prostate Cancer: A Retrospective Analysis. AJR Am J Roentgenol. 2022 Feb;218(2):333-340. doi: 10.2214/AJR.21.25961. Epub 2021 Aug 18. PMID 34406051

RESULTS

PARTICIPANT FLOW:
Groups:
- 68Ga-PSMA PET/MRI: Patients receive 68Ga-PSMA-11 IV. Patients then undergo PET/MRI after 45 minutes of administration of radiopharmaceutical injection.
  68Ga-PSMA-11: Undergo 68Ga-PSMA-11 PET/MRI Magnetic resonance imaging (MRI): Undergo 68Ga-PSMA-11 PET/MRI Positron Emission Tomography (PET): Undergo 68Ga-PSMA-11 PET/MRI
Period: Overall Study
Arm/Group | 68Ga-PSMA PET/MRI
Started | 74
Completed | 73
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | 68Ga-PSMA PET/MRI
Number analyzed (Participants) | 74
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 31
  >=65 years | 43
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 74
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 70
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 11
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 2
  White | 56
  More than one race | 0
  Unknown or Not Reported | 4
Region of Enrollment [Number; unit: participants]
  United States | 74

OUTCOME MEASURES:

1. Primary Outcome: 68Ga-PSMA-11 PET Detection of Prostate Cancer Metastasized to Lymph Nodes
Description: 68-gallium (68Ga)-prostate-specific membrane antigen (PSMA) positron emission tomography/magnetic resonance imaging (PET/MRI) will be used to detect regional nodal and distant metastases in participants with intermediate and high-risk prostate cancer scheduled to undergo prostatectomy with lymph node dissection. The data will be analyzed by imaging interpretation. Each participant will be interpreted as either positive or negative for the presence of metastatic disease by 68Ga-PSMA PET/MRI, as assessed by imaging interpretation. The outcome will be expressed as the number of participants with metastatic disease, as identified by PET/MRI, a number without dispersion.
Time Frame: 1 Day
Measure: Count of Participants; unit: Participants
Arm/Group | 68Ga-PSMA PET/MRI
Number analyzed (Participants) | 73
Participants | 19

2. Secondary Outcome: Histopathologic Detection of Prostate Cancer Metastasized to Lymph Nodes
Description: Participants that undergo prostatectomy will be evaluated for prostate cancer metastasis to the lymph nodes as determined by histopathology. Each participants will be interpreted as either positive or negative for the presence of metastatic disease by histopathology. The outcome will be expressed as the number of participants with metastatic disease, as identified by histopathology, a number without dispersion.
Time Frame: 1 Day
Population: Some participants elected to have alternatives to prostatectomy, such as external beam radiation or observation.
Measure: Count of Participants; unit: Participants
Arm/Group | 68Ga-PSMA PET/MRI
Number analyzed (Participants) | 64
Participants | 16

3. Secondary Outcome: Sensitivity of 68Ga-PSMA-11 PET/MRI
Description: 68-gallium (68Ga)-prostate-specific membrane antigen (PSMA) positron emission tomography/magnetic resonance imaging (PET/MRI) will be used to detect metastases in participants with intermediate and high-risk prostate cancer scheduled to undergo prostatectomy with lymph node dissection. For participants that undergo both procedures (68Ga-PSMA PET/MRI and prostatectomy), sensitivity of the 68Ga-PSMA PET/MRI detection of metastatic prostate cancer will be determined. For an individual participant, sensitivity means the 2 assessments are in agreement that the participant truly has (ie, true-positive) have the condition being tested for (ie, metastatic prostate cancer). The outcome is reported as the percentage of participants for which the 2 assessments are in agreement that metastatic prostate cancer is detected (true-positive), a number without dispersion.
Time Frame: 1 Day
Population: Some participants elected to have alternatives to prostatectomy, such as external beam radiation or observation.
Measure: Number; unit: Percentage of participants
Arm/Group | 68Ga-PSMA PET/MRI
Number analyzed (Participants) | 64
Percentage of participants | 56.2

4. Secondary Outcome: Specificity of 68Ga-PSMA-11 PET/MRI
Description: 68-gallium (68Ga)-prostate-specific membrane antigen (PSMA) positron emission tomography/magnetic resonance imaging (PET/MRI) will be used to detect metastases in participants with intermediate and high-risk prostate cancer scheduled to undergo prostatectomy with lymph node dissection. For participants that undergo both procedures (68Ga-PSMA PET/MRI and prostatectomy), specificity of the 68Ga-PSMA PET/MRI detection of metastatic prostate cancer will be determined. For an individual participant, specificity means the 2 assessments are in agreement that the participant does not (ie, true-negative) have the condition being tested for (ie, metastatic prostate cancer). The outcome is reported as the percentage of participants for which the 2 assessments are in agreement that metastatic prostate cancer is not detected (true-negative), a number without dispersion.
Time Frame: 1 Day
Population: Some participants elected to have alternatives to prostatectomy, such as external beam radiation or observation.
Measure: Number; unit: Percentage of participants
Arm/Group | 68Ga-PSMA PET/MRI
Number analyzed (Participants) | 64
Percentage of participants | 85.4

ADVERSE EVENTS:
Time Frame: up to 72 hours
Arm/Group | 68Ga-PSMA PET/MRI
All-Cause Mortality (participants affected / at risk) | 0/74
Serious Adverse Events (participants affected / at risk) | 0/74
Other Adverse Events (participants affected / at risk) | 0/74

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-08-28): https://cdn.clinicaltrials.gov/large-docs/51/NCT02678351/Prot_SAP_000.pdf
  • Informed Consent Form (2020-12-01): https://cdn.clinicaltrials.gov/large-docs/51/NCT02678351/ICF_001.pdf